CLINICAL TRIAL: NCT01222442
Title: A Single-centre, Randomised, Double-blind, Double-dummy, Placebo Controlled, 4-way Crossover Phase I Study to Investigate the Effect of 2 Single Doses (400 μg and 1200 µg) of Inhaled AZD3199 on QT/QTc Interval, Compared to Placebo, Using Moxifloxacin (Avelox®) as a Positive Control, in Healthy Male Volunteers
Brief Title: To Evaluate the Effect of AZD3199 on the Electrical Activity in the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Leonard Siew/Dr, Quintiles Drug Research Unit at Guy's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D0570C00004
Record Dates: First submitted 2010-10-12; First posted 2010-10-18 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Disease
Keywords: Respiratory disease; Bronchiolitis; Emphysema; Lung disease causing persistent narrowing of the airways
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiration Disorders; Bronchiolitis; Emphysema | interventions — AZD-3199; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): 400 µg AZD3199 + moxifloxacin placebo
  Interventions: Drug: AZD3199
- 2 (Experimental): 1200 µg AZD3199 + moxifloxacin placebo
  Interventions: Drug: AZD3199
- 3 (Active Comparator): AZD3199 placebo + moxifloxacin 400 mg
  Interventions: Drug: Moxifloxacin
- 4 (Placebo Comparator): AZD3199 placebo + moxifloxacin placebo
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Drug: AZD3199 — Single dose, oral inhalation
  Arms: 1; 2
Drug: Moxifloxacin — Single dose, oral encapsulated tablet
  Other Names: Avelox®
  Arms: 3
Other: Placebo comparator — Single dose, oral inhalation
  Arms: 4

SUMMARY:
The purpose of this research study is to evaluate the effect of AZD3199 on the electrical activity of the heart. The effect of AZD3199 will be compared to a licensed antibiotic (moxifloxacin). Moxifloxacin effects on the electrical activity of the heart are well known. Safety and tolerability of AZD3199 and how much AZD3199 enters the blood circulation will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years (inclusive)
* Have a body mass index (BMI) between 19 and 30 kg/m2 and a body weight between 60 and 100 kg.
* Be a non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start.
* Be able to inhale from the Turbuhaler inhaler according to given instructions.

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings at screening examination
* History of additional risk factors for Torsade de Pointes (eg, heart failure, hypokalaemia, or family history of long QT syndrome).
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of AZD3199 on the QT interval | Throughout the study
  QTcF or QTcI (algorithm based decision)

SECONDARY OUTCOMES:
To investigate the effect of AZD3199 on additional electrocardiogram variables | Throughout the study
  * QTcF or QTcI dependent on variable confirmed as primary
  * Holter-Bin QT
To assess the pharmacokinetics of single doses of AZD3199. | Throughout the study
  * AUC(0-24)
  * Cmax
  * tmax
To evaluate the safety and tolerability of single doses of AZD3199. | Throughout the study
  * Adverse events - type of events and number of subjects experiencing adverse events.
  * Laboratory safety assessments, pulse, blood pressure and electrocardiogram interpretation - Summarised using descriptive stats. Judged regarding high/low values or changes from pre-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&D, Lund, Sweden; Leonard Siew, MB CHB, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital, London
Locations (1):
- Research Site, London, UK, United Kingdom